CLINICAL TRIAL: NCT03847714
Title: Probiotics in Dementia
Acronym: PIDE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PIDE
Record Dates: First submitted 2019-02-11; First posted 2019-02-20 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2024-03

CONDITIONS: Dementia; Alzheimer, Mixed Type (Etiology)
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: similar looking and tasting placebo
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic (Active Comparator): Bifidobacterium bifidum W23, B. lactis W51, B. lactis W52, Lactobacillus acidophilus W22, L. casei W56, L. paracasei W20, L. plantarum W62, L. salivarius W24, Lactococcus lactis W19, 7.5 × 109 Colony Forming Units/g twice daily dissolved in water
  Interventions: Dietary Supplement: Omni-Biotic Stress Repair
- Placebo (Placebo Comparator): 3g of a similar looking and tasting powder, twice daily
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: Omni-Biotic Stress Repair — The probiotic supplement is a commercially available food for special medical purposes and includes 9 bacterial strains with at least 7.5 billion organisms (7.5 × 109 Colony Forming Units/g) per 1 portion (= 3 g).
  Other Names: Omni-Biotic SR-9, Winclove 825
  Arms: Probiotic
Dietary Supplement: placebo — similar looking and tasting powder
  Arms: Placebo

SUMMARY:
Dementia is associated with changes in gut microbiome composition, gut barrier dysfunction, intestinal inflammation and systemic inflammation. Probiotics are a possibility to modulate the gut-brain axis. In this study the effect of probiotics on the gut microbiome and, gut barrier function, inflammation and cognitive dysfunction will be studied.

DETAILED DESCRIPTION:
Dementia is a disease that presents with deterioration in memory, thinking, behaviour and the ability to perform everyday activities. Worldwide 47.5 million people are affected and incidence of dementia is increasing. Dementia leads to disability and dependency among older people worldwide and thereby has a huge physical, psychological, social and economic impact on caregivers, families and society. Alzheimer's disease (AD) is the most common form of dementia accounting for 60-70% of the cases; other forms include Lewy body dementia, frontotemporal dementia, vascular dementia and Parkinson's disease with dementia. In AD, pathologic protein aggregates of amyloid beta and hyperphosphorylated tangles of tau-protein which deposit as neurofibrillary tangles are typical features. This leads to neuroinflammation, mainly mediated by the innate immune system. The most important cells in this process are microglia cells, which represent the resident macrophages of the brain. Although microglia is able to remove extracellular amyloid beta, in later stages of the disease cells remain in a dystrophic state and cannot exert their beneficial functions. Microglia maturation and function is critically dependent on short-chain fatty acids produced by the gut microbiome and therefore highlights the microbiome as a potential diagnostic and therapeutic target in dementia.

The role of the commensal microbial population of the human body - especially the intestinal microbiome - in various diseases is emerging due to the development of advanced analysis techniques. Recently the concept of the gut brain-axis has been established. Several pathways including the autonomic nervous system, the enteric nervous system, the neuroendocrine system and the immune system allow a communication between gut and brain but may also be involved in disease development.

During ageing, the gut microbiome composition undergoes changes. A decrease in diversity, a loss of beneficial taxa and an increase of facultative pathogens has been described. Diet and the place of residence play an important role in the shaping of the microbiome. Aging is also associated with inflammation - often termed as "inflammaging" associated with an increase in gut permeability, mucosal inflammation and bacterial translocation.

Since the main risk factor for developing dementia, especially AD, is aging, it is very likely that the gut-brain axis is critically involved in dementia development.

Animal studies so far suggest that AD is associated with changes in the gut microbiome composition with a decrease in beneficial, anti-inflammatory genera. Furthermore, genetic alterations in amyloid genes can influence microbiome composition in mice, pointing towards a vicious cycle in AD development.

In humans, so far only limited evidence on the microbiome composition in patients with dementia is available. There is evidence that the composition of the microbiome in subgingival plaques is altered in dementia and associated with cognitive function. Recently the first human study identified phylum- through genus-wide differences in bacterial abundance including decreased Firmicutes, increased Bacteroidetes, and decreased Bifidobacterium in the stool of AD patients.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Dementia of Alzheimer type and mixed type (diagnosis by a board-certified neurologist/psychiatrist and according to ICD10)
* Mini Mental State Examination 21-26
* Stable treatment with anti-dementia drugs including phytotherapeutics (>3 months) or no intention to start anti-dementia drugs
* Informed consent

Exclusion Criteria:

* Other forms of dementia
* Inflammatory bowel diseases
* Liver cirrhosis
* Antibiotic treatment within the last 4 weeks
* Febrile illness within the last 4 weeks
* Acute hospital admission for dementia-unrelated reasons within the last 4 weeks
* Dysphagia
* Any other condition or circumstance, which, in the opinion of the investigator, would affect the patient's ability to participate in the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2019-06-15 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Butyrate producing bacteria | 6 months
  abundance of butyrate producing bacteria

SECONDARY OUTCOMES:
Butyrate producing bacteria | 12 months
  abundance of butyrate producing bacteria
diaminooxidase concentration in serum | 6 months
  marker of intestinal permeability
diaminooxidase concentration in serum | 12 months
  marker of intestinal permeability
zonulin concentration in stool | 6 months
  marker of intestinal permeability
zonulin concentration in stool | 12 months
  marker of intestinal permeability
calprotectin concentration in stool | 6 months
  marker of intestinal inflammation
calprotectin concentration in stool | 12 months
  marker of intestinal inflammation
soluble CD 14 concentration in serum | 6 months
  marker of systemic inflammation
soluble CD 14 concentration in serum | 12 months
  marker of systemic inflammation
lipopolysaccharide binding protein concentration in serum | 6 months
  marker of systemic inflammation
lipopolysaccharide binding protein concentration in serum | 12 months
  marker of systemic inflammation
lipopolysaccharide concentration in serum | 6 months
  marker of bacterial translocation
lipopolysaccharide concentration in serum | 12 months
  marker of bacterial translocation
peptidoglycan concentration in serum | 6 months
  marker of bacterial translocation
peptidoglycan concentration in serum | 12 months
  marker of bacterial translocation
bacterial DNA concentration in serum | 6 months
  marker of bacterial translocation
bacterial DNA concentration in serum | 12 months
  marker of bacterial translocation
Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS cog) | 6 months
  Questionnaire to assess cognitive function, 0-70 points
Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS cog) | 12 months
  Questionnaire to assess cognitive function, 0-70 points
Mini mental state examination | 6 months
  Questionnaire to assess cognitive function, 0-30 points
Mini mental state examination | 12 months
  Questionnaire to assess cognitive function, 0-30 points
clinician's interview-based impression of change with caregiver input (CIBIC+) | 6 months
  Questionnaire to assess overall change during the study, 1-7 points
clinician's interview-based impression of change with caregiver input (CIBIC+) | 12 months
  Questionnaire to assess overall change during the study, 1-7 points
Barthel index | 6 months
  Assessment of activities of daily living, 0-100 points
Barthel index | 12 months
  Assessment of activities of daily living, 0-100 points

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University Graz, Graz, Austria

IPD SHARING:
Plan to Share IPD: Yes
microbiome sequencing data will be published at nucleotide archive
Supporting Information: Study Protocol
Time Frame: at time of publication; no limit
Access Criteria: open